CLINICAL TRIAL: NCT01976767
Title: Protocol for the European Multi-Centre Study Understanding Severe Asthma Longitudinal Assessment of Adults With Severe Asthma
Brief Title: Longitudinal Assessment of Adults With Severe Asthma
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. P.J. Sterk, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 10/H0721/66
Record Dates: First submitted 2013-10-22; First posted 2013-11-06 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Asthma
Keywords: Sputum; Clinical cohorts; Smokers; Asthma; Biopsies; Severe asthma; Collaborative research; Phenotyping; Lipidomics; Transcriptomics; Proteomics; Paediatric cohort; Systems Biology
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cohort A: Adults: severe asthmatics on high dose ICS and / or OCS
- Cohort B: Adults: current smokers or ex-smokers, severe asthmatics on high dose ICS and / or OCS
- Cohort C: Adults: non-smokers, mild to moderate asthmatics on regular inhaled corticosteroids (ICS)
- Cohort D: Adults: healthy volunteers, non-smokers, non-asthmatic with pre bronchodilator FEV1 > 80% predicted

SUMMARY:
Cross-sectional study to characterize cohorts of subjects with asthma and healthy controls in terms of clinical features, physiological measurements and non-invasive measurement of biomarkers and develop phenotype handprints for adults with severe asthma

ELIGIBILITY:
General Inclusion Criteria:

1. Able to give written informed consent prior to participation in the study, which includes ability to comply with the requirements and restrictions listed in the consent form. Informed consent must be obtained prior to undertaking any study procedures.
2. Male or female subject aged 18 years or older at screening.
3. Able to complete the study and all measurements.
4. Able to read, comprehend, and write at a sufficient level to complete study related materials.
5. Subjects will be allowed to enrol in other studies while taking part on this study. However, Permission from the Scientific Board must be obtained to enrol or allow the continued participation of a subject enrolled in another study.

General Exclusion Criteria:

1. As a result of medical interview, physical examination or screening investigation the physician responsible considers the subject unfit for the study either because of the risk to the subject due to the study or the influence this may have on the study results.
2. The subject has a history of recreational drug use or other allergy, which, in the opinion of the responsible physician, contra-indicates their participation.
3. Subject is female who is pregnant or lactating or up to 6 weeks post partum or 6 weeks cessation of breast feeding. If a woman is subsequently found to have been pregnant at the time of an assessment data from that assessment will not be included in the analyses.
4. The subject has participated within 3 months of the first dose in a study using a new molecular entity, or the first dose in any other study investigating drugs or having participated within three months in a study with invasive procedures. Any U-BIOPRED assessments should be deferred until 3 months after the first dose or invasive procedure. Permission from the Scientific Board must be obtained to enroll or allow the continued participation of a subject enrolled in another study.
5. Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures.
6. The subject has a recent history of incapacitating psychiatric disorders
7. History or current evidence of an upper or lower respiratory infection or symptoms (including common cold) within 2 weeks of baseline assessments (assessments should be deferred).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Severe asthma cohorts: uncontrolled asthma symptoms or frequent severe exacerbations
  * Mild-moderate asthma cohorts: controlled or partially controlled asthma symptoms
  * Healthy controls: non-asthmatic healthy individuals free of significant disease
Sampling Method: Non-Probability Sample
Enrollment: 725 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbations | 3 years
  Number, duration and severity of exacerbations over the time of the study
Lung function decline over the course of the study | 3 years
Changes in asthma medication | 3 years
  in particular ICS dose, over the duration of the study
Daily symptoms and short acting beta agonist (SABA) usage | 3 years
  measured during the telemonitoring study
Asthma control questionnaire (ACQ) at baseline and changes over the course of the study | 3 years
Upper airway symptoms as assessed by the sino-nasal outcomes test (SNOT) at baseline and changes over the course of the study | 3 years
Sleep and daytime drowsiness as assessed by the Epworth sleepiness scale at baseline and changes over the course of the study | 3 years
Measurement of pulmonary function including spirometry, plethysmography, bronchodilator reversibility and respiratory impedance by forced oscillation technique | 3 years
Radiological parameters such as computerized tomography (CT) scan, including assessment of lung structure | 3 years
Measurement of inflammatory cell counts in blood, sputum and bronchoalveolar lavage (BAL) | 3 years
Histopathology of bronchial biopsies in a sub group of subjects | 3 years
  immunohistochemistry for inflammatory cells and matrix remodelling
Transcriptomics, proteomics and metabolomics will be used on samples such as blood, urine and endobronchial biopsies | 3 years
  to develop clinically useful phenotype handprints
Quality of life as assessed by the asthma quality of life questionnaire (AQLQ) | 3 years
Anxiety and depression as assessed by the hospital anxiety and depression scale (HADS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sterk, Dr., Principal Investigator — Academic Medical Centre University of Amsterdam, The Netherlands; Ratko Djukanovic, Dr., Principal Investigator — Southampton General Hospital, UK; Stephen Fowler, Dr., Principal Investigator — Respiratory Research Group, Education and Research Centre, Wythenshawe Hospital, UK; Kian Fan Chung, Dr., Principal Investigator — Imperial College London, UK; Barbro Dahlén, Dr., Principal Investigator — Karolinska Institutet; Andrew Szczeklik, Dr., Principal Investigator — Uniwersytet Jagielloński - Collegium Medicum, Kraków, Poland; Thomas Geiser, Dr., Principal Investigator — Inselspital and University of Bern, Switzerland; Ildiko Horvath, Dr., Principal Investigator — University School of Medicine, Budapest, Hundary; Pascal Chanez, Dr., Principal Investigator — Université de la Méditerranee, Marseille, France; Jens Hohlfeld, Dr., Principal Investigator — Fraunhofer Institute for Toxicology and Experimental Medicine, Hannover; Thomas Sandström, Dr., Principal Investigator — Department of Public Health and Clinical Medicine, Division of Medicine, Umea, Sweden; Dominick Shaw, Dr., Principal Investigator — Nottingham City Hospita, Nottingham, UK; Per Sigvald Bakke, Dr., Principal Investigator — Haukeland University Hospital, Bergen, Norway; Riccardo Polosa, Dr., Principal Investigator — Policlinico Vittorio Emmanuele, Catania, Italy; Paolo Montuschi, Dr., Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS

REFERENCES:
- [Derived] Reinke SN, Naz S, Chaleckis R, Gallart-Ayala H, Kolmert J, Kermani NZ, Tiotiu A, Broadhurst DI, Lundqvist A, Olsson H, Strom M, Wheelock AM, Gomez C, Ericsson M, Sousa AR, Riley JH, Bates S, Scholfield J, Loza M, Baribaud F, Bakke PS, Caruso M, Chanez P, Fowler SJ, Geiser T, Howarth P, Horvath I, Krug N, Montuschi P, Behndig A, Singer F, Musial J, Shaw DE, Dahlen B, Hu S, Lasky-Su J, Sterk PJ, Chung KF, Djukanovic R, Dahlen SE, Adcock IM, Wheelock CE; U-BIOPRED Study Group. Urinary metabotype of severe asthma evidences decreased carnitine metabolism independent of oral corticosteroid treatment in the U-BIOPRED study. Eur Respir J. 2022 Jun 30;59(6):2101733. doi: 10.1183/13993003.01733-2021. Print 2022 Jun. PMID 34824054
- [Derived] Kolmert J, Gomez C, Balgoma D, Sjodin M, Bood J, Konradsen JR, Ericsson M, Thorngren JO, James A, Mikus M, Sousa AR, Riley JH, Bates S, Bakke PS, Pandis I, Caruso M, Chanez P, Fowler SJ, Geiser T, Howarth P, Horvath I, Krug N, Montuschi P, Sanak M, Behndig A, Shaw DE, Knowles RG, Holweg CTJ, Wheelock AM, Dahlen B, Nordlund B, Alving K, Hedlin G, Chung KF, Adcock IM, Sterk PJ, Djukanovic R, Dahlen SE, Wheelock CE; U-BIOPRED Study Group, on behalf of the U-BIOPRED Study Group. Urinary Leukotriene E4 and Prostaglandin D2 Metabolites Increase in Adult and Childhood Severe Asthma Characterized by Type 2 Inflammation. A Clinical Observational Study. Am J Respir Crit Care Med. 2021 Jan 1;203(1):37-53. doi: 10.1164/rccm.201909-1869OC. PMID 32667261
- [Derived] Emma R, Bansal AT, Kolmert J, Wheelock CE, Dahlen SE, Loza MJ, De Meulder B, Lefaudeux D, Auffray C, Dahlen B, Bakke PS, Chanez P, Fowler SJ, Horvath I, Montuschi P, Krug N, Sanak M, Sandstrom T, Shaw DE, Fleming LJ, Djukanovic R, Howarth PH, Singer F, Sousa AR, Sterk PJ, Corfield J, Pandis I, Chung KF, Adcock IM, Lutter R, Fabbella L, Caruso M; U-BIOPRED Study Group. Enhanced oxidative stress in smoking and ex-smoking severe asthma in the U-BIOPRED cohort. PLoS One. 2018 Sep 21;13(9):e0203874. doi: 10.1371/journal.pone.0203874. eCollection 2018. PMID 30240401